CLINICAL TRIAL: NCT04611009
Title: Treatment Effect and Relevance on Daily Life of a Video-supervised Sensorimotor Training Program and Its Influence on the Pathophysiology in Writer's Cramp
Brief Title: Video-supervised Motor and Awareness Training in Writer's Cramp
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DE 579/17
Record Dates: First submitted 2020-06-10; First posted 2020-11-02 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Writer's Cramp
Keywords: dystonia; training; kinematic writing analysis; COPM; functional magnetic resonance imaging
MeSH Terms: conditions — Dystonic Disorders; Dystonia

STUDY DESIGN:
Intervention Model Description: randomized, controlled, double blinded trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded towards their participation in the two arms Clinical scales, kinematic writing anlysis and functional MRI will be analyzed by persons, who are blinded to the type of training group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motor training (Experimental): intervention: motor training
  Interventions: Behavioral: motor training
- awareness training (Active Comparator): intervention: mindfulness exercises
  Interventions: Behavioral: mindfulness exercises

INTERVENTIONS:
Behavioral: motor training — In the sensorimotor training program task-specific and non-task specific aspects will be combined. It will start with assignments to improve general finger and wrist movements. After four weeks more specific writing exercises will be added.
  Arms: motor training
Behavioral: mindfulness exercises — The awareness training will contain mindfulness exercises. The goal is to consciously experience the here and now in sensual perception of oneself and the environment.
  Arms: awareness training

SUMMARY:
Writer's cramp is the most common task-specific dystonia. It is characterized by involuntary co-contraction of antagonistic muscles during writing. This disabling condition may force patients to give up their occupation. In this study the efficacy of a twelve months long-term training in patients with writer's cramp will be investigated. Two different programs will be offered: The first one will consist of a sensorimotor, the second one of an awareness training. All patients will benefit from video-based supervision with the aim to establish a practice-oriented therapeutic approach that will be available to all patients independently of their home location. The treatment effect will be measured primary with the patient-centered Canadian Occupational Performance Measure (COPM) and secondary with clinical scales to assess the clinical efficacy and everyday constraints. Writing will be assessed with a computer-based kinematic writing analysis. To evaluate the influence on the brain network, several functional magnetic resonance imaging (fMRI) evaluations will be performed. This project is of minimal risk without negative side effects from the training. The risks for the MRI experiment are equal to a non-contrast standard MRI investigation.

ELIGIBILITY:
Inclusion Criteria:

* Right handed idiopathic WC according to standardized criteria (simple and complex WC, any dystonic posture (including flexion, extension, pronation, supination))
* able to participate in video-calls

Exclusion Criteria:

* Additional neurological or psychiatric diseases
* left-handed patients
* last botulinum toxin treatment <3 months, remaining weakness from the last injection
* concomitant use of anticholinergics or sedating medication

Exclusion criteria for MRI:

* Cardiac pacemaker, electronic or metal implants
* pregnancy or suspected pregnancy
* severe ametropia, anxiety in small rooms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Change from baseline to month 4, 8, 12
  The Canadian Occupational Performance Measure will serve as the primary outcome measure. Patients grade their self-perceived performance and satisfaction of writing related occupations in daily life in respect to the goals they had identified and prioritized. The COPM ist patient centered end reflects the real life of the participants.

SECONDARY OUTCOMES:
kinematic writing analysis | Change from baseline to month 4, 8, 12
  The kinematic handwriting analysis will be performed on a pressure sensitive digitizing tablet, that is connected to a laptop to measure movements of the pencil during writing. Regularity of writing will be calculated from this data. All subjects will write a standardized sentence and draw superimposed circles to characterize handwriting movements.
Writer's Cramp Rating Scale | Change from baseline to month 4, 8, 12
  The video based Writer's Cramp Rating Scale will serve as a secondary outcome parameter. The videos are rated by a blinded movement disorder specialist according to flexion / extension of arm / wrist / fingers during writing.
writing during functional magnetic resonance imaging (fMRI) | Change from baseline to month 4, 8, 12
  During this task participants will be instructed to a) write a sentence using an MR-compatible tablet and b) imagine writing in randomized order. The task is performed during a fMRI measurement. With the imaginary task artefacts are avoided and activation during movement planning will be investigated in the fMRI.
qualitative interviews | Change from baseline to month 4, 12
  The purpose of the semi-structured qualitative interviews about the training procedures is to optimize the training and to differentiate between responders and non-responders. The interviews will be will be transcribed word-for-word and analyzed using the qualitative content analysis.
Arm Dystonia Disability Scale | Change from baseline to month 4, 8, 12
  The Arm Dystonia Disability Scale will be applied to assess how dystonia interferes with manual activities during daily life (writing, buttoning, hygiene, eating, job or household).
Serial Reaction Time Task during functional magnetic resonance imaging (fMRI) | Change from baseline to month 4, 8, 12
  The Serial Reaction Time Task is a standardized method to investigate motor sequence learning and to induce cerebellar activation. We expect that abnormal cerebellar activity in patients compared to controls normalizes after training.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten E Zeuner, Prof. MD, Principal Investigator — Kiel University
Locations (1):
- Kiel University, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Baur B, et.al. Effects of modified pen grip and handwriting training on writer's cramp. Arch Phys Med Rehabil 2009;90(5):867-875. — http://pubmed.ncbi.nlm.nih.gov/19406309/
- See also: Bleton JP, Vidailhet M, Bourdain F, Ducorps A, Schwartz D, et al. Somatosensory cortical remodelling after rehabilitation and clinical benefit of in writer's cramp. J Neurol Neurosurg Psychiatry 2011;82(5):574-577. — http://pubmed.ncbi.nlm.nih.gov/20562399/
- See also: Castrop F, Dresel C, Hennenlotter A, Zimmer C, Haslinger B. Basal ganglia-premotor dysfunction during movement imagination in writer's cramp. Mov Disord 2012;27(11):1432-1439. — http://pubmed.ncbi.nlm.nih.gov/22328061/
- See also: Delnooz CC, Helmich RC, Medendorp WP, Van de Warrenburg BP, Toni I. Writer's cramp: increased dorsal premotor activity during intended writing. Hum Brain Mapp 2013;34(3):613-625. — http://pubmed.ncbi.nlm.nih.gov/22113948/
- See also: Gallea C, Horovitz SG, Najee-Ullah M, Hallett M. Impairment of a parieto-premotor network specialized for handwriting in writer's cramp. Hum Brain Mapp 2016;37(12):4363-4375. — http://pubmed.ncbi.nlm.nih.gov/27466043/
- See also: Granert O, Peller M, Gaser C, Groppa S, Hallett M, Knutzen A, Deuschl G, Zeuner KE, Siebner HR. Manual activity shapes structure and function in contralateral human motor hand area. Neuroimage 2011;54(1):32-41. — http://pubmed.ncbi.nlm.nih.gov/20708692/
- See also: Hallett M. Pathophysiology of writer's cramp. Hum Mov Sci 2006;25(4-5):454-463. — http://pubmed.ncbi.nlm.nih.gov/16859794/
- See also: Planton S, Longcamp M, Peran P, Demonet JF, Jucla M. How specialized are writing-specific brain regions? An fMRI study of writing, drawing and oral spelling. Cortex 2017;88:66-80. — http://pubmed.ncbi.nlm.nih.gov/28081451/
- See also: Rothkirch I, Granert O, Knutzen A, Wolff S, et al. Dynamic causal modeling revealed dysfunctional effective connectivity in both, the cortico-basal-ganglia and the cerebello-cortical motor network in writers' cramp. Neuroimage Clin 2018;18:149-159. — http://pubmed.ncbi.nlm.nih.gov/29868443/
- See also: Shakkottai VG, Batla A, Bhatia K , Dauer WT, Dresel C, et al. Current Opinions and Areas of Consensus on the Role of the Cerebellum in Dystonia. Cerebellum 2017;16(2):577-594. — http://pubmed.ncbi.nlm.nih.gov/27734238/
- See also: Stahl CM, Frucht SJ. Focal task specific dystonia: a review and update. J Neurol 2017;264(7):1536-1541. — http://pubmed.ncbi.nlm.nih.gov/28039522/
- See also: Zeuner KE, Shill HA, Sohn YH, Molloy FM, Thornton BC, Dambrosia JM, Hallett M. Motor training as treatment in focal hand dystonia. Mov Disord 2005;20(3):335-341. — http://pubmed.ncbi.nlm.nih.gov/15486996/
- See also: Zeuner KE, Peller M, Knutzen A, et al. How to assess motor impairment in writer's cramp. Mov Disord 2007;22(8):1102-1109. — http://pubmed.ncbi.nlm.nih.gov/17230462/
- See also: Zeuner KE, Molloy FM. Abnormal reorganization in focal hand dystonia-sensory and motor training programs to retrain cortical function. NeuroRehabilitation 2008;23(1):43-53. — http://pubmed.ncbi.nlm.nih.gov/18356588/
- See also: Zeuner KE, Peller M, Knutzen A, Hallett M, Deuschl G, Siebner HR. Motor re-training does not need to be task specific to improve writer's cramp. Mov Disord 2008;23(16):2319-2327. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4149415/
- See also: Zeuner KE, Knutzen A, Granert O, et al. Increased volume and impaired function: the role of the basal ganglia in writer's cramp. Brain Behav 2015;5(2):e00301. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4309880/